CLINICAL TRIAL: NCT05743803
Title: Observance of Preoperative Fasting Time a Before-and-after Sensitization Campaign to Preoperative Fasting Guidelines Study
Brief Title: Observance of Preoperative Fasting Time a Before-and-after Sensitization Campaign to Fasting Guidelines Study
Acronym: BreakFast
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-AR23_00060
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Fasting
Keywords: fasting; quality of recovery; surgery
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before: This group will undergo their preoperative fasting period as standard care.
- After: This group will undergo their preoperative fasting period after the sensitization campaign about preoperative fasting rules.
  Interventions: Other: Sensititization campaign on preoperative fasting rules

INTERVENTIONS:
Other: Sensititization campaign on preoperative fasting rules — * Planned and repeated mandatory on site lecture about pre-operative guidelines for surgeons, anesthetists and paramedics.
  * Reminder display in surgical wards and consults.
  * Individualized fasting cards for patients.
  * Short message service reminder on pre-operative fasting rules for patients.
  * Medical fasting prescription with clear fasting times.
  Groups: After

SUMMARY:
The goal of this before and after observational study is to evaluate the impact of a global sensitization campaign (targeted on surgeons, anesthetist and patients) about pre-operative fasting in an adult population. The main questions it aims to answer are:

* Does the sensitization campaign reduce fasting time?
* Does reduce fasting time increase quality of post-operative recovery?

Sensitization campaign will be performed between the before and after phases, it will include:

* Planned and repeated mandatory on site lecture about pre-operative guidelines for surgeons, anesthetists and paramedics.
* Reminder display in surgical wards and consults.
* Individualized fasting cards for patients.
* Short message service reminder on pre-operative fasting rules for patients.
* Medical fasting prescription with clear fasting times.

ELIGIBILITY:
Inclusion Criteria:

- Adult undergoing a surgical procedure.

Exclusion Criteria:

* Already intubated patient before surgery.
* Redo surgery during the same hospitalization
* Medical indication of fasting (e.g : occlusive syndrome)
* Patient unable to anwser the questionnaire.
* Patient under lawful protection
* Pregnant women
* Minor (<18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing a surgical procedure (scheduled or urgent) at the CHU d'Angers (France) during the inclusion period.
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Fasting time | Before surgery
  Liquid and solid fasting time before surgery (minutes)

SECONDARY OUTCOMES:
Preoperative oral carbohydrate loading | 2 hours preoperative period
  Rate of oral cardbohydrate intake in the 2 hours preoperative period (percentage)
Fasting exceeding 12 hours | Before surgery
  Rate of fasting duration superior to 12 hours (liquid or solid) (percentage)
Preoperative anxiety | Before surgery
  Scale of preoperative anxiety from 0 (no anxiety) to 10 (maximum anxiety possible)
Preoperative discomfort | Before surgery
  Scale of preoperative disomfort from 0 (no discomfort) to 10 (maximum discomfort possible)
Feeling of thirst | Before surgery
  Qualitative scale of preoperative thirst (none, moderate, significant)
Feeling of hunger | Before surgery
  Qualitative scale of preoperative hunger (none, moderate, significant)
Preoperative nausea or vomiting | Before surgery
  Rate of nausea or vomit in the preoperative period (percentage)
Rate of postoperative nausea or vomiting | Day of surgery
  Rate of nausea or vomit during the post-operative period (percentage)
Patient satisfaction toward communication and explanation about preoperative fasting. | Day of surgery
  Binary answer (yes or no)
Post-operative quality of recovery | Day 1 after surgery
  French Quality of Recovery 15 score (
Length of stay | Maximum 30 days follow up
  Length of stay (days)
Post-operative surgical complication | Maximum 30 days follow up
  Clavien-dindo classification from 0 (no complication) to 5 (death)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No